CLINICAL TRIAL: NCT05173909
Title: Effects of BIS Closed Loop Target Controlled Infusion on Perioperative Inflammatory Response and Prognosis of Elderly Patients Undergoing Laparoscopic Radical Gastrectomy for Gastric Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhonghua Chen,MD (Other)
Responsible Party: Sponsor-Investigator, Zhonghua Chen,MD, Head of anesthesiology, Shaoxing Hospital of Zhejiang University
Organization: Shaoxing Hospital of Zhejiang University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 032
Record Dates: First submitted 2021-12-15; First posted 2021-12-30 (Actual); Last update posted 2021-12-30 (Actual); Status verified 2021-12

CONDITIONS: The Effect of BIS Closed-loop Target Control on Postoperative Operation
Keywords: BIS closed-loop target controlled infusion; sedation deep; laparoscopic radical gastrectomy; elderly patients

STUDY DESIGN:
Intervention Model Description: A total of 73 patients were selected and divided into two groups according to random number table method: BIS closed loop target controlled infusion group with BIS value of 55 (group H) and BIS closed loop-target controlled infusion group with BIS value of 45 (group L), The final grouping results were 36 cases in group H and 37 cases in group L. All enrolled patients signed informed consent forms.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: None of the participants，care providers and outcomes assessors knew the grouping, and only the experimenter had to adjust BIS. In this way, the description of the treatment effects and adverse reactions of the subjects, as well as the recording of the experimenter's various reactions, can be as objective as possible.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group H (Experimental): BIS closed-loop target controlled infusion group with BIS value of 55
  Interventions: Device: BIS closed-loop target controlled infusion
- group L (Experimental): BIS closed-loop target controlled infusion group with BIS value of 45
  Interventions: Device: BIS closed-loop target controlled infusion

INTERVENTIONS:
Device: BIS closed-loop target controlled infusion — BIS was monitored by connecting the BIS monitor (BISXP, Aspects Medical Systems, USA). The corresponding value was set on the BIS detector and connected to the targy-controlled infusion pump to automatically adjust the plasma drug concentration of propofol

SUMMARY:
The purpose of this study is to find the elderly patients with laparoscopic gastric cancer radical is suitable the BIS closed round target control level of anesthesia depth of sedation, can decrease the elderly laparoscopic gastric cancer radical surgery in patients with perioperative inflammatory reaction, and reduce the incidence of perioperative pulmonary complications such as, for elderly patients with gastric cancer radical perioperative inflammation control to provide the reference and provide guidance for clinical anesthesia work.

DETAILED DESCRIPTION:
In this study, elderly patients undergoing laparoscopic radical gastrectomy for gastric cancer were randomly divided into BIS closed circle target controlled infusion (BIS) 55 group and 45 group, and the levels of perioperative inflammatory response indicators IL-6, TNF-α and IL-10 at different depths of anesthesia and sedation were recorded. The duration of stay in anesthesia recovery room, quality of recovery, postoperative pain and postoperative pulmonary complications were observed. Objective To evaluate the feasibility of BIS closed loop target controlled infusion in elderly patients undergoing laparoscopic radical gastrectomy for gastric cancer.

Perioperative period is a process of intense stress response, which is mainly manifested by the production and aggregation of inflammatory factors, which adversely affect multiple organs such as brain, heart and lung, and is an important risk factor for increasing postoperative complications and postoperative mortality .

Perioperative inflammatory response status has a clear relationship with postoperative recovery of patients, and perioperative anesthesia and sedation depth management and precision anesthesia is one of the most critical links to control the stress response, and appropriate anesthesia and sedation depth control and stress regulation can significantly improve the prognosis of patients . How to reduce the adverse effects of perioperative stress response on patients has been the focus of research and attention in recent years.

ELIGIBILITY:
Inclusion Criteria:

Age 65 or above ASA-PSTYPE I or II Both male and female Laparoscopic radical gastrectomy for gastric cancer

Exclusion Criteria:

The patient had abnormal liver, kidney and other important organs before surgery The patient has chronic pain Patients with neurological or mental disorders Long-term use of sedation, painkillers and antipsychotic drugs The patient has contraindications for opioid use

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 73 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Postoperative complications | Within one week after surgery
  pulmonary infection, oxygenation injury, arrhythmia, bleeding, intestinal paralysis, incision infection, renal insufficiency, cognitive dysfunction, etc.
mortality rate | Within 30 days after surgery
  mortality rate
Serum LEVELS of IL-2, IL-4, IL-6, IL-10, TNF-ɑ, IFN-γ | Within three days of the surgery
  Serum levels of IL-2, IL-4, IL-6, IL-10, TNF-ɑ and IFN-γ were determined immediately before operation, 2 hours after operation, 24 hours after operation and 72 hours after operation

CONTACTS AND LOCATIONS:
Locations (1):
- Shaoxing People's Hospital, Shaoxing, China

IPD SHARING:
Plan to Share IPD: No